CLINICAL TRIAL: NCT04093323
Title: A Phase II Study of Type-1 Polarized Dendritic Cell (aDC1) -Based Treatment in Combination With Tumor-Selective Chemokine Modulation (CKM: Interferon Alpha 2b, Rintatolimod and Celecoxib) in Melanoma Patients With Primary PD-1/PD-L1 Resistance
Brief Title: Polarized Dendritic Cell (aDC1) Based Treatment, Interferon Alpha-2, Rintatolimod, and Celecoxib for the Treatment of HLA-A2+ Refractory Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding completed
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 82419; NCI-2019-05911 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 82419 (Other: Roswell Park Cancer Institute); P01CA234212 (NIH)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: HLA-A2 Positive Cells Present; Refractory Melanoma
MeSH Terms: conditions — Melanoma | interventions — Celecoxib; Immune Checkpoint Inhibitors; Introns; Interferon alpha-2; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (IFNA2, rintatolimod, celecoxib, alphaDC1 cell based treatment) (Experimental): Patients receive recombinant interferon alpha-2 IV over 30 minutes, rintatolimod IV over 2.5 hours, and celecoxib PO BID on days 1-3. Beginning cycle 2, patients also receive alpha-type-1 polarized dendritic cells ID on day 1. Treatment repeats every 3 weeks up to 4 cycles in the absence of disease progression or unacceptable toxicity. At 12 weeks, patients with progressive disease may switch to ipilimumab with or without a PD-1/PD-L1 inhibitor and patients with a complete response CR, PR, or stable disease SD may switch to a PD-1/PD-L1 inhibitor or best alternative care.
  Interventions: Biological: Alpha-type-1 Polarized Dendritic Cells; Drug: Celecoxib; Drug: PD-1 Ligand Inhibitor; Drug: PD1 Inhibitor; Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod

INTERVENTIONS:
Biological: Alpha-type-1 Polarized Dendritic Cells — Given ID
  Other Names: alphaDC1
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
Drug: PD-1 Ligand Inhibitor — Given IV
  Other Names: PD-1 Ligands Inhibitor
Drug: PD1 Inhibitor — Given IV
  Other Names: PD-1 Inhibitor; Programmed Cell Death Protein 1 Inhibitor; Protein PD-1 Inhibitor
Biological: Recombinant Interferon Alfa-2b — Given IV
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen

SUMMARY:
This phase II trial studies how well polarized dendritic cell (aDC1) based therapy, interferon alpha-2, rintatolimod, and celecoxib work together in treating patients with HLA-A2 positive (+) melanoma that has not responded to previous treatment (refractory). The aDC1 cell-based treatment contains white blood cells (dendritic cells or DCs) that stimulates the immune system. Interferon alpha-2 can improve the body's natural response to infections and other diseases. It can also interfere with the division of cancer cells and slow tumor growth. Rintalolimid may stimulate the immune system. Celecoxib is a drug that reduces pain. This study is being done to find out if the combination of the study cell-based treatment (aDC1 dendritic cells) and interferon alpha-2, rintatolimod, and celecoxib can prevent the growth and/or progression of melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the objective response rate to treatment with an autologous alpha-type-1 polarized dendritic cells (alphaDC1)/TBVA cell-based treatment (alpha-type-1-polarized dendritic cells loaded with tumor blood vessel-targeting antigenic peptides) plus cytokine modulating (CKM) regimen (rintatolimod, recombinant interferon alpha-2 [IFN-alpha2b] and, celecoxib) in human leukocyte antigen (HLA)-A2+ subjects with primary PD-1 resistant immuno-oncology (IO)-refractory melanoma (who will continue the original PD-1/PD-L1 regimen for 12 weeks).

SECONDARY OBJECTIVES:

I. To evaluate the immune-related objective response rate (objective response rate [ORR]; per immune-related Response Evaluation Criteria in Solid Tumors [iRECIST];) in the above patient population treated with autologous alphaDC1/TBVA cell-based treatment plus cytokine CKM regimen followed by continued treatment with PD-1/PD-LI blockade (+/- CTLA4 blockade or LAG3 blockade).

II. Evaluate rate of durable responses (> 6 months) on the combination treatment in the above patient population treated with autologous alphaDC1/TBVA cell-based treatment plus cytokine CKM regimen followed by continued treatment with PD-1/PD-L1 blockade (+/- CTLA4 blockade or LAG3 blockade).

EXPLORATORY OBJECTIVES:

I. Examine whether the combination of peptide-loaded autologous alphaDC1 cell-based treatment and tumor-selective chemokine modulation (CKM: IFN-a2b, rintatolimod, and celecoxib) improves the overall survival (OS) and immune-related progression-free survival (iPFS) in HLA-A2+ subjects PD-1/PD-L1-refractory melanoma compared to the historical control of the best supportive care.

II. Identify the intratumoral and systemic immune correlates of the response to treatment.

OUTLINE:

Patients receive recombinant interferon alpha-2 intravenously (IV) over 30 minutes, rintatolimod IV over 2.5 hours, and celecoxib orally (PO) twice daily (BID) on days 1-3. Beginning cycle 2, patients also receive alpha-type-1 polarized dendritic cells intradermally (ID) on day 1. Treatment repeats every 3 weeks up to 4 cycles in the absence of disease progression or unacceptable toxicity. At 12 weeks, patients with progressive disease may switch to ipilimumab with or without a PD-1/PD-L1 inhibitor and patients with a complete response (CR), partial response (PR), or stable disease (SD) may switch to a PD-1/PD-L1 inhibitor or best alternative care.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be HLA-A2+. Retesting is not required for patients who have previous documented positivity
* Have IO-refractory melanoma with primary PD-1/PD-L1resistance. Note: Any lines of prior therapies are allowed, but the last line needs to include an anti PD-1 or anti PD-L1 agent. The prior treatments may include any standard and/or experimental therapies
* Have >= 1 tumor site amenable to core needle biopsy that is not the site of disease used to measure antitumor response
* Have measurable disease based on RECIST 1.1 criteria present
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Platelets >= 75,000/microliter
* Hemoglobin >= 9 g/deciliter
* Absolute neutrophil count (ANC) >= 1500/microliter
* Creatinine < 1.5 x institutional upper limit of normal (ULN) OR creatinine clearance >= 50 mL/min by Cockcroft-Gault formula for subjects with creatinine levels >= 1.5 x ULN
* Total bilirubin not greater than 1.5 x institutional ULN, except for patients with known Gilbert's Syndrome, who are eligible to no more than 2 x institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) no greater than 3 x institutional ULN OR, no greater than 5 x ULN for subjects with liver metastases
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Candidate for continuation/resumption of anti-PD-1/PD-L1 blockade (in parallel to DC vaccine and CKM)

Exclusion Criteria:

* Is currently being treated with systemic immunosuppressive agents, including steroids: Subjects will be ineligible until 3 weeks after removal from immunosuppressive treatments, except when they are administered as replacement therapy for endocrine dysfunction (and receive no more than 10 mg prednisone or equivalent: inhaled steroids are allowed)
* Has had prior anti-cancer therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., no more than grade 1 or at baseline) from adverse events due to a previously administered agent, except for neuropathy (no more than grade 2) or alopecia or vitiligo (any grade)
* Has a known additional malignancy that is progressing or requires active treatment
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Treated brain metastases are allowed, if stable for more than 4 weeks (and receive no more than 10 mg prednisone or equivalent: inhaled steroids are allowed).
* Has a history of cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia (within 3 months of signing consent) or, subject has a New York Heart Association classification of III or IV
* Has an active infection requiring systemic therapy
* Has known active hepatitis B or hepatitis C infection
* Has known immunosuppressive disease (e.g. human immunodeficiency virus [HIV], acquired immunodeficiency syndrome [AIDS] or other immune depressing disease). Testing is not mandatory
* Has known serious hypersensitivity reactions to pegylated (peg)-interferon alpha-2b or interferon alpha-2b
* Prior allergic reaction or hypersensitivity to sulfonamides, celecoxib, or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Has received a blood transfusion in the two weeks prior to leukapheresis
* Women of child bearing potential who are pregnant or nursing
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate or unacceptable risk to receive study drug regimen
* Patients who showed initial response to PD-1/PD-L1 blockade and developed secondary resistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At 12 weeks
  Will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Will be carried out by an exact binomial test of a proportion within a Simon two-stage design.

SECONDARY OUTCOMES:
ORR | At 6 months
  Will be evaluated using immune-related RECIST (iRECIST) criteria in patients that continue on with either PD1 and/or CTLA4 blockade after meeting the 12-week primary objective treated with autologous alpha-type-1 polarized dendritic cells (alphaDC1)/tumor blood vessel-targeting antigenic peptides (TBVA) cell-based treatment plus cytokine modulating (CKM) regimen followed by re-treatment with PD1 blockade (+/- CTLA4 blockade). The analysis will be primarily descriptive and consist of sample proportions and the corresponding 95% confidence intervals.
Durable objective response rate (>= 6 months) | From time of first confirmed response assessed up to 2 years
  Will be evaluated on patients treated autologous alphaDC1/TBVA cell-based treatment plus cytokine CKM regimen followed by retreatment with PD1 blockade (+/- CTLA4 blockade). The analysis will be primarily descriptive and consist of sample proportions and the corresponding 95% confidence intervals.

OTHER OUTCOMES:
Immune-related progressive free survival | Up to 2 years
  Will be evaluated using iRECIST criteria. Will be compared to the historical control of the best supportive care and to identify the intratumoral and systemic immune correlates of the response to treatment. Will be analyzed by a Cox regression model as a function of various biomarker combinations.
Overall survival | Up to 2 years
  Will be compared to the historical control of the best supportive care and to identify the intratumoral and systemic immune correlates of the response to treatment. Will be analyzed by a Cox regression model as a function of various biomarker combinations.
Change in density of CD8 positive cytotoxic T cells | Baseline up to week 11
  Will be evaluated using the OmniSeq immune report card (IRC). Will be analyzed by a Cox regression model as a function of various biomarker combinations.
Change in density of molecular biomarkers | Baseline up to week 11
  Will be evaluated using the OmniSeq IRC. Will be analyzed by a Cox regression model as a function of various biomarker combinations.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Puzanov, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT04093323/ICF_000.pdf